CLINICAL TRIAL: NCT00179049
Title: Evaluation of Immunoregulatory Cells in Hematopoietic Stem Cell Transplant (HSCT)
Brief Title: Evaluation of Immunoregulatory Cells in Hematopoietic Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Adetola A. Kassim, MD, Vanderbilt University
Other Study IDs: BMT 030261
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-12-15 (Estimated); Status verified 2008-12

CONDITIONS: Hematopoietic Stem Cell Transplantation; Graft vs Host Disease
Keywords: T-Lymphocyte Subsets
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators' hypothesis is that the graft-versus-tumor effect can be enhanced while minimizing the complications of graft-versus-host disease.

DETAILED DESCRIPTION:
The investigators' hypothesis is that the graft-versus-tumor effect can be enhanced while minimizing the complications of graft-versus-host disease (GVHD) by determining the qualitative and quantitative changes in T regulatory cells throughout the transplant process. Their understanding of this can lead to new treatment strategies and improved clinical therapeutic implications.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-70 years old undergoing either autologous transplant or allogeneic transplant for various hematologic conditions

Exclusion Criteria:

* Patients < 18 or > 70 years old undergoing either autologous transplant or allogeneic transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18-70 years old undergoing either autologous transplant or allogeneic transplant for various hematologic conditions
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2003-04; Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adetola A Kassim, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States